CLINICAL TRIAL: NCT00848770
Title: Manipulation of Arterial Pressure Early in Non Thrombolysed Acute Ischemic Stroke: Effects on Death and Neurological Disability
Brief Title: Manipulation of Arterial Pressure in Acute Ischemic Stroke
Acronym: MAPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Hospital de Clinicas de Porto Alegre, GPPG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPA 07-470
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-02

CONDITIONS: Stroke, Acute
Keywords: Stroke, Acute; Systolic Pressure of Blood
MeSH Terms: conditions — Stroke | interventions — esmolol; Norepinephrine; Nucleolus Organizer Region

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1, 140 to 160 mmHg (Active Comparator): Esmolol, NPS or NOR
  Interventions: Drug: Esmolol, Sodium Nitroprussiate (NPS) or Norepinephrine (NOR); Drug: Esmolol, NPS or NOR; Drug: manipulation of SAP
- 2, 161 to 180 mmHg (Active Comparator): Esmolol, NPS or NOR
  Interventions: Drug: Esmolol, Sodium Nitroprussiate (NPS) or Norepinephrine (NOR); Drug: Esmolol, NPS or NOR; Drug: manipulation of SAP
- 3, 181 to 200 mmHg (Active Comparator): Esmolol, NPS or NOR
  Interventions: Drug: Esmolol, Sodium Nitroprussiate (NPS) or Norepinephrine (NOR); Drug: Esmolol, NPS or NOR; Drug: manipulation of SAP

INTERVENTIONS:
Drug: Esmolol, Sodium Nitroprussiate (NPS) or Norepinephrine (NOR) — Esmolol(2,5g /10ml + SG5% 240ml = 10mg/ml). Start with a bolus of 500mcg/kg in 1 min (ou 0,5mg/kg)and maintain the dose of 50mcg/kg/min (or 0,05mg/kg/min). Increase de infusion in 25mcg/kg/min after each 5 min until the randomized SAP or if the heart beat is lower than 60. The maximum dose is 200ug/kg/min (ou 0,2 mg/kg/min). If the randomized SAP do not reach the goal pressure with the maximum dose of esmolol, start a infusion of sodium nitroprussiate (NPS).
  NPS (50mg + SG5% 250ml= 200mcg/ml). No bolus. Start the infusion with 0,2 mcg/kg/min and maintain 0,5 a 5mcg/kg/min. Increase de dose each 15 min to a maximum of 10mcg/kg/min.
  NOR: (8mg/8ml + SG5% 242ml=32mcg/ml)No bolus. Start 1 to 5 mcg/min to a maximum dose of 20mcg/min.
  Other Names: Esmolol, NPS or NOR
Drug: Esmolol, NPS or NOR — We use one of the three drug to manipulate the systolic arterial pressure
Drug: manipulation of SAP — Esmolol or NPS or NOR
  Other Names: Esmolol or NPS or NOR

SUMMARY:
This is a controlled clinical trial among non thrombolysed acute ischemic stroke patients to determine the effects of three levels of arterial pressure on death and neurological disability. After the admission in the vascular unit of the Emergency Department the patients are randomized to maintain during the first 24h the Systolic Arterial Pressure in tree levels of pressure: 140 to 160 mmHg; 161 to 180 mmHg and 181 to 200 mmHg. The end point of the study is the Modified Rankin score and mortality in three month after the discharge.

DETAILED DESCRIPTION:
To maintain the tree levels of systolic arterial pressure during de first 24h we will use one of the two strategies:1) infusion of 500 to 1000ml of saline solution and/or norepinephrine solution to increase de systolic pressure or 2) infusion of esmolol or nitroprussiate solution to decrease de pressure. Every patient will have a transcranial doppler study in the first 24h to measure the mean velocity of cerebral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older, with the first Acute Ischemic Stroke within the first 6 hours of the symptoms and not candidate to thrombolysis
* We will also include patients with previous Ischemic Stroke with Ranking score 0 or 1

Exclusion Criteria:

* Improuvment of the symptoms rapidly (in the first 15 min after admission)
* Seizures not related do the acute ischemic stroke
* Previous ischemic stroke in the last 6 weeks and with Ranking score > 1
* Haemorrhagic stroke
* Anticoagulation
* Hypoglycemia
* Shock
* Acute heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Ranking score and mortality | Three month

CONTACTS AND LOCATIONS:
Overall Officials: Luiz A Nasi, Physician, Principal Investigator — Hospital de Clínicas de Porto Alegre / UFRGS
Locations (1):
- Hospital de Clínicas de Porto Alegre/ UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Potter J, Robinson T, Ford G, James M, Jenkins D, Mistri A, Bulpitt C, Drummond A, Jagger C, Knight J, Markus H, Beevers G, Dewey M, Lees K, Moore A, Paul S; CHHIPS Trial Group. CHHIPS (Controlling Hypertension and Hypotension Immediately Post-Stroke) Pilot Trial: rationale and design. J Hypertens. 2005 Mar;23(3):649-55. doi: 10.1097/01.hjh.0000160224.94220.e7. PMID 15716709
- See also: Clinical trial of Manipulation of Arterial Pressure Early in Acute Ischemic Stroke — http://clinicaltrials.gov/ct2/show/NCT00848770